CLINICAL TRIAL: NCT04085913
Title: Intraoperative Injection of Exparel Effect on Postoperative Opioid Use in Thyroid and Parathyroid Surgery
Brief Title: Exparel Injection Effect on Postoperative Opioid Usage
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Tabitha L. Galloway, Assistant Professor of Clinical Otolaryngology, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014881
Record Dates: First submitted 2019-06-21; First posted 2019-09-11 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Thyroid; Parathyroid Adenoma
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, randomized research study to evaluate postoperative pain medication usage in patients scheduled and receiving thyroid/parathyroid surgery. Patients will be randomized into three different study groups, each receiving a different regiment of treatment.
Who Masked: Participant
Masking Description: During the consenting process, participants will be informed about the randomization aspect of the study. However, they will not be told what category/group they will be randomized into. To help with the randomization, the study team will enter the needed patient information into www.randomizer.org, which will categorize the patients into the desired groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Current Practice (Active Comparator): Thyroid or parathyroid surgery with local injection of lidocaine and epinephrine preincision, as is current practice.
  Interventions: Drug: Lidocaine Epinephrine
- Bupivicaine HCL (Experimental): Thyroid or parathyroid surgery with local injection of bupivicaine HCL and Epinephrine preincision.
  Interventions: Drug: Bupivacaine Hydrochloride-EPINEPHrine
- Exparel Injection (Experimental): Thyroid and parathyroid surgery with local injection of lidocaine and epinephrine preincison and Exparel postincision
  Interventions: Drug: Lidocaine Epinephrine, Bupivacaine Hydrochloride-EPINEPHrine

INTERVENTIONS:
Drug: Lidocaine Epinephrine — Preincision injection, as is current practice
  Arms: Current Practice
Drug: Bupivacaine Hydrochloride-EPINEPHrine — Preincision injection
  Other Names: Exparel
  Arms: Bupivicaine HCL
Drug: Lidocaine Epinephrine, Bupivacaine Hydrochloride-EPINEPHrine — Preincison injection of lidocaine and epinephrine and a postincision injection of Exparel
  Other Names: Exparel
  Arms: Exparel Injection

SUMMARY:
The question proposed by this study, is one of patient outcomes. Does intraoperative injection of Exparel decrease postoperative use of opioid pain medications in patients undergoing thyroid and parathyroid surgery? The trial seeks to assess the effect that Exparel has on postoperative pain control.

DETAILED DESCRIPTION:
Patients will be identified in clinic as good candidates for surgical intervention based on current standard of care. Once participants are consented, they will be randomly placed into one of three categories. The first category being patients undergoing surgery with local injection of lidocaine and epinephrine as is current practice. The second category of patients will undergo surgery with local injection of bupivacaine HCL and epinephrine preincision. The third group will undergo surgery with local injection of lidocaine and epinephrine preincision and Exparel postincision. As stated above, all patients will undergo surgery as planned, which will be standard of care, with the exception of the local anesthetic and timing of the injection. Postoperatively, patient's pain scores and opioid usage will be evaluated. Patients will be monitored by either using the patient's electronic medical record or by a pain journal that will be provided to the patients. The patients will record their pain using a scale of 1-10 with the FACES scale, as well as medication usage. Patients will return to their first postoperative appointment to further discuss their pain levels as well as medication usage. An ANOVA test will be used to determine if there is a significant difference in the amount of opioids taken postoperatively, in oral morphine equivalents, between these three groups. Opioid usage will then be compared between participants in different categories of local anesthetic to determine if there is an effect of postoperative opioid usage between different anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years Patients requiring parathyroid/thyroid surgery based on the standard of care English as primary language

Exclusion Criteria:

* Patients under the age of 18 years Patients with previous history of opioid abuse Patients with a true allergy to any local anesthetic Patients with a true allergy to any opioid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of opioid use when given Exparel intraoperatively | After surgery, patients will be monitored for two weeks, until they return for their first postoperative appointment.
  Utilizing pain scale daily diary, we will evaluate the incidence of opioid usage in patients that have undergone thyroid/parathyroid surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tabitha Galloway, MD, Principal Investigator — University of Missouri Department of Otolaryngology-Head and Neck Surgery
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan, because IPD will not be shared with other researchers.